CLINICAL TRIAL: NCT00981058
Title: A Randomized, Multicenter, Open-Label Phase 3 Study of Gemcitabine-Cisplatin Chemotherapy Plus Necitumumab (IMC-11F8) Versus Gemcitabine-Cisplatin Chemotherapy Alone in the First-Line Treatment of Patients With Stage IV Squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: First-line Treatment of Participants With Stage IV Squamous Non-Small Cell Lung Cancer With Necitumumab and Gemcitabine-Cisplatin
Acronym: SQUIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Parexel (Industry); PPD Development, LP (Industry); Medidata Solutions (Industry); Laboratory Corporation of America (Industry); University of Colorado, Denver (Other); Thermo Fisher Scientific FS (Other); ICON Clinical Research (Industry); Pacific Biomarkers (Other); Sysmex Inostics GmbH (Industry); Intertek (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13909; CP11-0806 (Other: ImClone Systems); I4X-IE-JFCC (Other: Eli Lilly and Company); 2009-013838-25 (EudraCT Number)
Record Dates: First submitted 2009-09-18; First posted 2009-09-22 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2025-06-18 (Actual); Status verified 2025-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Squamous; Non Small Cell Lung Cancer; First line treatment; Monoclonal; Antibodies; Epidermal Growth Factor Receptor (EGFR)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — necitumumab; Gemcitabine; LY2334737; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Necitumumab + Gemcitabine + Cisplatin (Experimental): Necitumumab: 800 milligrams (mg) I.V. infusion on Days 1 and 8 of every 3 week cycle.
  Continues until progressive disease, toxicity, noncompliance, or withdrawal.
  Gemcitabine: 1250 milligrams/square meter (mg/m2) on Days 1 and 8 of every 3 week cycle.
  Continues for a maximum of six cycles.
  Cisplatin: 75 mg/m2 IV on Day 1 of every 3 week cycle. Continues for a maximum of six cycles.
  Interventions: Biological: Necitumumab; Drug: Gemcitabine; Drug: Cisplatin
- Gemcitabine + Cisplatin (Active Comparator): Gemcitabine: 1250 mg/m2 on Days 1 and 8 of every 3 week cycle. Continues for a maximum of six cycles.
  Cisplatin: 75 mg/m2 IV on Day 1 of every 3 week cycle. Continues for a maximum of six cycles.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Biological: Necitumumab — Administered intravenously.
  Continues until progressive disease, toxicity, noncompliance, or withdrawal.
  Other Names: IMC-11F8; LY3012211
  Arms: Necitumumab + Gemcitabine + Cisplatin
Drug: Gemcitabine — Administered intravenously.
  Continues for a maximum of six cycles.
  Other Names: LY2334737
Drug: Cisplatin — Administered intravenously.
  Continues for a maximum of six cycles.

SUMMARY:
The research study is testing the investigational drug necitumumab (IMC-11F8) in the treatment of advanced non-small cell lung cancer. The aim of this study is to determine if necitumumab, given together with a standard chemotherapy combination consisting of cisplatin and gemcitabine will be more effective in improving participant disease than the standard chemotherapy combination alone.

DETAILED DESCRIPTION:
Multinational, randomized, multicenter, open-label, Phase III study of 1093 participants (age ≥ 18 years) with histologically- or cytologically-confirmed, stage IV squamous-cell NSCLC, who have received no prior therapy for metastatic disease, will be randomized on a 1:1 basis to receive first-line necitumumab plus chemotherapy consisting of gemcitabine and cisplatin in study Arm A, or gemcitabine-cisplatin chemotherapy alone in study Arm B. Baseline radiographic assessment of disease will be performed within 21 days prior to randomization (first treatment will be administered within 7 days following randomization). Participants will undergo radiographic assessment of disease status (computed tomography or magnetic resonance imaging) every 6 weeks (± 3 days), until there is radiographic documentation of progressive disease (PD). Chemotherapy will continue for a maximum of six cycles in each arm (or until there is radiographic documentation of PD, toxicity requiring cessation, protocol noncompliance or withdrawal of consent); participants in Arm A only will continue to receive necitumumab until there is radiographic documentation of PD, toxicity requiring cessation, protocol noncompliance, or withdrawal of consent.

After the end-of-study-visit (following PD), follow-up information regarding further anticancer treatment and survival will be collected every 2 months (± 7 days). For participants who discontinue study for reasons other than PD (eg, symptomatic deterioration), information on disease progression will also be collected until PD is documented. Follow-up will continue as long as the participant is alive, or until the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed squamous NSCLC
* Has Stage IV disease at the time of study entry
* Measurable or nonmeasurable disease at the time of study entry as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.0) (participants with only truly nonmeasurable disease are not eligible)
* Has resolution to Grade ≤ 1 of all clinically significant toxic effects of prior chemotherapy, surgery, radiotherapy, or hormonal therapy (with the exception of alopecia)
* Has adequate hepatic function
* Has adequate renal function
* Has adequate hematologic function
* If female, is surgically sterile, postmenopausal, or compliant with a highly effective contraceptive method (failure rate < 1%) during and for 6 months after the treatment period (oral hormonal contraception alone is not considered highly effective and must be used in combination with a barrier method)
* If male, the participant is surgically sterile or compliant with a highly effective contraceptive regimen during and for 6 months after the treatment period
* Female participants of childbearing potential must have a negative serum pregnancy test within 7 days prior to randomization
* Has archived tumor tissue available for analysis of EGFR and KRAS mutation status (by PCR) and EGFR gene copy number (by FISH); minimum of four slides, paraffin-embedded tissue, required

Exclusion Criteria:

* Has nonsquamous NSCLC (adenocarcinoma/large cell or other)
* Has received prior anticancer therapy with monoclonal antibodies, signal transduction inhibitors, or any therapies targeting the EGFR, vascular endothelial growth factor (VEGF), or VEGF receptor
* Has received previous chemotherapy for advanced NSCLC (participants who have received adjuvant chemotherapy are eligible if the last administration of the prior adjuvant regimen occurred at least 1 year prior to randomization)
* Has undergone major surgery or received any investigational therapy in the 4 weeks prior to randomization
* Has undergone chest irradiation within 12 weeks prior to randomization (except palliative irradiation of bone lesions, which is allowed)
* Has brain metastases that are symptomatic or require ongoing treatment with steroids or anticonvulsants. Participants who have undergone previous radiotherapy for brain metastases, who are now nonsymptomatic and no longer require treatment with steroids or anticonvulsants, are eligible
* Has superior vena cava syndrome contraindicating hydration
* Has current clinically-relevant coronary artery disease or uncontrolled congestive heart failure
* Has experienced myocardial infarction within 6 months prior to randomization
* Has an ongoing or active infection (requiring antibiotics), including active tuberculosis or known infection with the human immunodeficiency virus
* Has a history of significant neurological or psychiatric disorders, including dementia, seizures, or bipolar disorder
* Has any National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 3.0 Grade ≥ 2 peripheral neuropathy
* Has significant third space fluid retention, requiring repeated drainage
* Has any other serious uncontrolled medical disorders or psychological conditions that would, in the opinion of the investigator, limit the participant's ability to complete the study or sign an informed consent document
* Has a known allergy / history of hypersensitivity reaction to any of the treatment components, including any ingredient used in the formulation of necitumumab (IMC-11F8), or any other contraindication to one of the administered treatments
* Is pregnant or breastfeeding
* Has a known history of drug abuse
* Has a concurrent active malignancy other than adequately-treated basal cell carcinoma of the skin or preinvasive carcinoma of the cervix. A participant with previous history of malignancy other than NSCLC is eligible, provided that he/she has been free of disease for ≥ 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1093 (Actual)
Dates: Start 2010-01-07 (Actual); Primary Completion 2013-06-17 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (160):
- United States (15):
  - ImClone Investigational Site, Chandler, Arizona
  - ImClone Investigational Site, Fayetteville, Arkansas
  - ImClone Investigational Site, Sacramento, California
  - ImClone Investigational Site, Galesburg, Illinois
  - ImClone Investigational Site, Goshen, Indiana
  - ImClone Investigational Site, Wichita, Kansas
  - ImClone Investigational Site, Hazard, Kentucky
  - ImClone Investigational Site, Baltimore, Maryland
  - ImClone Investigational Site, Jefferson City, Missouri
  - ImClone Investigational Site, Lincoln, Nebraska
  - ImClone Investigational Site, New York, New York
  - ImClone Investigational Site, Akron, Ohio
  - ImClone Investigational Site, Camp Hill, Pennsylvania
  - ImClone Investigational Site, Memphis, Tennessee
  - ImClone Investigational Site, Fairfax, Virginia
- Australia (5):
  - ImClone Investigational Site, Garran, New South Wales
  - ImClone Investigational Site, Westmead, New South Wales
  - ImClone Investigational Site, Wollongong, New South Wales
  - ImClone Investigational Site, East Bentleigh, Victoria
  - ImClone Investigational Site, Geelong, Victoria
- Austria (2):
  - ImClone Investigational Site, Linz
  - ImClone Investigational Site, Vienna
- Belgium (3):
  - ImClone Investigational Site, Duffel
  - ImClone Investigational Site, Liège
  - ImClone Investigational Site, Namur
- Brazil (11):
  - ImClone Investigational Site, Barretos
  - ImClone Investigational Site, Brasilia, Distrito Federal
  - ImClone Investigational Site, Goiânia
  - ImClone Investigational Site, Ijuí
  - ImClone Investigational Site, Itajaí
  - ImClone Investigational Site, Lajeado
  - ImClone Investigational Site, Porto Alegre/RS
  - ImClone Investigational Site, Salvador
  - ImClone Investigational Site, Santo André
  - ImClone Investigational Site, São Paulo
  - ImClone Investigational Site, São Paulo - SP
- Canada (3):
  - ImClone Investigational Site, Saint John, New Brunswick
  - ImClone Investigational Site, Brampton, Ontario
  - ImClone Investigational Site, Saskatoon, Saskatchewan
- Croatia (3):
  - ImClone Investigational Site, Dubrovnik
  - ImClone Investigational Site, Pula
  - ImClone Investigational site, Zagreb
- France (12):
  - ImClone Investigational Site, Brest
  - ImClone Investigational Site, Caen
  - ImClone Investigational Site, Draguignan
  - ImClone Investigational Site, Grenoble
  - ImClone Investigational Site, Le Mans
  - ImClone Investigational Site, Lille
  - ImClone Investigational Site, Lyon
  - ImClone Investigational Site, Marseille
  - ImClone Investigational Site, Paris
  - ImClone Investigational Site, Rennes
  - ImClone Investigational Site, Saint-Jean
  - ImClone Investigational Site, Toulon Armées
- Germany (17):
  - ImClone Investigational Site, Berlin
  - ImClone Investigational Site, Essen
  - ImClone Investigational Site, Frankfurt
  - ImClone Investigational Site, Gauting
  - ImClone Investigational Site, Großhansdorf
  - ImClone Investigational Site, Halle
  - ImClone Investigational Site, Hamburg
  - ImClone Investigational Site, Heidelberg
  - ImClone Investigational Site, Hemer
  - ImClone Investigational Site, Hofheim
  - ImClone Investigational Site, Karlsruhe
  - ImClone Investigational Site, Lostau
  - ImClone Investigational Site, Löwenstein
  - ImClone Investigational Site, München
  - ImClone Investigational Site, Münster
  - ImClone Investigational Site, Regensburg
  - ImClone Investigational Site, Ulm
- Greece (4):
  - ImClone Investigational Site, Athens
  - ImClone Investigational Site, Heraklion, Crete
  - ImClone Investigational Site, Pátrai
  - ImClone Investigational Site, Thessaloniki
- Hungary (7):
  - ImClone Investigational Site, Budapest
  - ImClone Investigational Site, Deszk
  - ImClone Investigational Site, Farkasgyepü
  - ImClone Investigational Site, Mosonmagyaróvár
  - ImClone Investigational Site, Székesfehérvár
  - ImClone Investigational Site, Szombathely
  - ImClone Investigational Site, Törökbálint
- Italy (8):
  - ImClone Investigational Site, Lido di Camaiore, Lucca
  - ImClone Investigational Site, Aviano, Pordenone
  - ImClone Investigational Site, Frosinone
  - ImClone Investigational Site, Genova
  - ImClone Investigational Site, Milan
  - ImClone Investigational Site, Monza
  - ImClone Investigational Site, Parma
  - ImClone Investigational Site, Perugia
- Philippines (6):
  - ImClone Investigational Site, Cebu
  - ImClone Investigational Site, Cebu City
  - ImClone Investigational Site, Davao City
  - ImClone Investigational Site, Makati City
  - ImClone Investigational Site, Manila
  - ImClone Investigational Site, Quezon City
- Poland (8):
  - ImClone Investigational Site, Olsztyn
  - ImClone Investigational Site, Otwock
  - ImClone Investigational Site, Poznan
  - ImClone Investigational Site, Radom
  - ImClone Investigational Site, Rzeszów
  - ImClone Investigational Site, Szczecin
  - ImClone Investigational Site, Torun
  - ImClone Investigational Site, Wroclaw
- Portugal (3):
  - ImClone Investigational Site, Coimbra
  - ImClone Investigational Site, Lisbon
  - ImClone Investigational Site, Porto
- Romania (7):
  - ImClone Investigational Site, Brasov
  - ImClone Investigational Site, Bucharest
  - ImClone Investigational Site, Cluj-Napoca
  - ImClone Investigational Site, Craiova, Dolj
  - ImClone Investigational Site, Iași
  - ImClone Investigational Site, Piatra Neamţ
  - ImClone Investigational Site, Sibiu
- Russia (9):
  - ImClone Investigational Site, Ivanovo
  - ImClone Investigational Site, Kirov
  - ImClone Investigational Site, Krasnodar
  - ImClone Investigational Site, Moscow
  - ImClone Investigational Site, Omsk
  - ImClone Investigational Site, Saint Petersburg
  - ImClone Investigational Site, Smolensk
  - ImClone Investigational Site, Ufa
  - ImClone Investigational Site, Yaroslavl
- Serbia (4):
  - ImClone Investigational Site, Belgrade
  - ImClone Investigational Site, Kamenitz
  - ImClone Investigational Site, Kragujevac
  - ImClone Investigational Site, Niš
- ImClone Investigational Site, Singapore, Singapore
- Slovakia (3):
  - ImClone Investigational Site, Bratislava
  - ImClone Investigational Site, Nitra
  - ImClone Investigational Site, Poprad
- South Africa (3):
  - ImClone Investigational Site, Bloemfontein, Free State
  - ImClone Investigational Site, Pretoria, Gauteng
  - ImClone Investigational Site, Durban, KwaZulu-Natal
- South Korea (5):
  - ImClone Investigational Site, Incheon
  - ImClone Investigational Site, Jeonju
  - ImClone Investigational Site, Seongnam
  - ImClone Investigational Site, Seoul
  - ImClone Investigational Site, Suwon
- Spain (9):
  - ImClone Investigational Site, Seville, Andalusia
  - ImClone Investigational Site, Ávila, Castille and León
  - ImClone Investigational Site, Barcelona, Catalonia
  - ImClone Investigational Site, Terrassa, Catalonia
  - ImClone Investigational Site, Madrid, Communidad de Madrid
  - ImClone Investigational Site, Majadahonda, Communidad de Madrid
  - ImClone Investigational Site, Barcelona
  - ImClone Investigational Site, L'Hospitalet de Llobregat
  - ImClone Investigational Site, Madrid
- ImClone Investigational Site, Taichung, Taiwan
- Thailand (2):
  - ImClone Investigational Site, Chiang Mai
  - ImClone Investigational Site, Songkhla
- United Kingdom (9):
  - ImClone Investigational Site, Aberdeen
  - ImClone Investigational Site, Bournemouth
  - ImClone Investigational Site, Dundee
  - ImClone Investigational Site, Edinburgh
  - ImClone Investigational Site, Guildford
  - ImClone Investigational Site, Liverpool
  - ImClone Investigational Site, London
  - ImClone Investigational Site, Manchester
  - ImClone Investigational Site, Preston

REFERENCES:
- [Derived] Ciuleanu T, Socinski MA, Obasaju C, Luft AV, Szczesna A, Szafranski W, Ramlau R, Balint B, Molinier O, Depenbrock H, Nanda S, Paz-Ares L, Thatcher N. Efficacy and Safety of Necitumumab Continuation Therapy in the Phase III SQUIRE Study of Patients With Stage IV Squamous Non-Small-Cell Lung Cancer. Clin Lung Cancer. 2018 Mar;19(2):130-138.e2. doi: 10.1016/j.cllc.2017.10.004. Epub 2017 Oct 13. PMID 29158123
- [Derived] Paz-Ares L, Socinski MA, Shahidi J, Hozak RR, Soldatenkova V, Kurek R, Varella-Garcia M, Thatcher N, Hirsch FR. Correlation of EGFR-expression with safety and efficacy outcomes in SQUIRE: a randomized, multicenter, open-label, phase III study of gemcitabine-cisplatin plus necitumumab versus gemcitabine-cisplatin alone in the first-line treatment of patients with stage IV squamous non-small-cell lung cancer. Ann Oncol. 2016 Aug;27(8):1573-9. doi: 10.1093/annonc/mdw214. Epub 2016 May 20. PMID 27207107
- [Derived] Reck M, Socinski MA, Luft A, Szczesna A, Dediu M, Ramlau R, Losonczy G, Molinier O, Schumann C, Gralla RJ, Bonomi P, Brown J, Soldatenkova V, Chouaki N, Obasaju C, Peterson P, Thatcher N. The Effect of Necitumumab in Combination with Gemcitabine plus Cisplatin on Tolerability and on Quality of Life: Results from the Phase 3 SQUIRE Trial. J Thorac Oncol. 2016 Jun;11(6):808-18. doi: 10.1016/j.jtho.2016.03.002. Epub 2016 Mar 12. PMID 26980471
- [Derived] Thatcher N, Hirsch FR, Luft AV, Szczesna A, Ciuleanu TE, Dediu M, Ramlau R, Galiulin RK, Balint B, Losonczy G, Kazarnowicz A, Park K, Schumann C, Reck M, Depenbrock H, Nanda S, Kruljac-Letunic A, Kurek R, Paz-Ares L, Socinski MA; SQUIRE Investigators. Necitumumab plus gemcitabine and cisplatin versus gemcitabine and cisplatin alone as first-line therapy in patients with stage IV squamous non-small-cell lung cancer (SQUIRE): an open-label, randomised, controlled phase 3 trial. Lancet Oncol. 2015 Jul;16(7):763-74. doi: 10.1016/S1470-2045(15)00021-2. Epub 2015 Jun 1. PMID 26045340

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers are defined as those participants who died due to any cause in this study.
Groups:
- Necitumumab + Gemcitabine + Cisplatin: Necitumumab + Gemcitabine + Cisplatin
  Necitumumab: 800 milligrams (mg) I.V. infusion on Days 1 and 8 of every 3 week cycle.
  Continues until progressive disease, toxicity, noncompliance, or withdrawal.
  Gemcitabine: 1250 milligrams/square meter (mg/m2) on Days 1 and 8 of every 3 week cycle.
  Continues for a maximum of six cycles.
  Cisplatin: 75 mg/m2 IV on Day 1 of every 3 week cycle.
  Continues for a maximum of six cycles.
- Gemcitabine + Cisplatin: Gemcitabine + Cisplatin
  Gemcitabine: 1250 mg/m2 on Days 1 and 8 of every 3 week cycle.
  Continues for a maximum of six cycles.
  Cisplatin: 75 mg/m2 IV on Day 1 of every 3 week cycle.
  Continues for a maximum of six cycles.
Period: Overall Study
Arm/Group | Necitumumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin
Started | 545 | 548
Received at Least 1 Dose of Study Drug | 538 | 541
Completed | 476 | 487
Not Completed | 69 | 61
Not completed — Progressive Disease | 38 | 31
Not completed — Lost to Follow-up | 3 | 2
Not completed — Physician Decision | 4 | 5
Not completed — Randomization Error | 0 | 1
Not completed — Withdrawal by Subject | 24 | 22

BASELINE CHARACTERISTICS:
Groups:
- Necitumumab + Gemcitabine + Cisplatin: Necitumumab + Gemcitabine + Cisplatin
  Necitumumab: 800 mg I.V. infusion on Days 1 and 8 of every 3 week cycle.
  Continues until progressive disease, toxicity, noncompliance, or withdrawal.
  Gemcitabine: 1250 mg/m2 on Days 1 and 8 of every 3 week cycle.
  Continues for a maximum of six cycles.
  Cisplatin: 75 mg/m2 IV on Day 1 of every 3 week cycle.
  Continues for a maximum of six cycles.
- Total: Total of all reporting groups
Arm/Group | Necitumumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin | Total
Number analyzed (Participants) | 545 | 548 | 1093
Age, Continuous [Median (Full Range); unit: years] | 62.0 [32 to 84] | 62.0 [32 to 86] | 62.0 [32 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 90 | 185
  Male | 450 | 458 | 908
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 56 | 111
  Not Hispanic or Latino | 489 | 490 | 979
  Unknown or Not Reported | 1 | 2 | 3
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 43 | 42 | 85
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 6 | 11
  White | 457 | 456 | 913
  More than one race | 1 | 0 | 1
  Other | 38 | 43 | 81
Region of Enrollment [Number; unit: participants]
  Russian Federation | 94 | 101 | 195
  Singapore | 1 | 2 | 3
  United States | 20 | 16 | 36
  Thailand | 3 | 6 | 9
  Portugal | 8 | 9 | 17
  Greece | 18 | 14 | 32
  Austria | 4 | 4 | 8
  Brazil | 28 | 30 | 58
  Korea, Republic of | 24 | 23 | 47
  Poland | 69 | 59 | 128
  Slovakia | 9 | 10 | 19
  France | 34 | 39 | 73
  Serbia | 11 | 13 | 24
  Croatia | 2 | 4 | 6
  Romania | 46 | 45 | 91
  Hungary | 43 | 41 | 84
  Philippines | 12 | 8 | 20
  United Kingdom | 9 | 10 | 19
  Spain | 33 | 25 | 58
  Canada | 2 | 4 | 6
  Belgium | 4 | 4 | 8
  Taiwan | 3 | 2 | 5
  Italy | 13 | 12 | 25
  South Africa | 2 | 2 | 4
  Australia | 4 | 6 | 10
  Germany | 49 | 59 | 108
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) at Baseline [Number; unit: participants] — ECOG classifies participants according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death). 1 participant with ECOG PS 3 was randomized to the Gemcitabine + Cisplatin arm but did not receive treatment.
  participants
    0 | 164 | 180 | 344
    1 | 332 | 320 | 652
    2 | 49 | 47 | 96
    3 | 0 | 1 | 1
Smoking History [Number; unit: participants]
  Ex-Light Smoker | 18 | 26 | 44
  Non-Smoker | 26 | 27 | 53
  Smoker | 500 | 495 | 995
  Missing | 1 | 0 | 1
Disease Stage at Study Entry [Number; unit: participants] — Stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body). Stage IIIB - the cancer has spread to nearby tissue or spread to far away lymph nodes. Stage IV - the cancer has spread to other organs of the body such as the other lung, brain, or liver.
  participants
    Stage IIIB | 1 | 1 | 2
    Stage IV | 543 | 546 | 1089
    Missing | 1 | 1 | 2
Disease Histology [Number; unit: participants]
  Squamous | 543 | 545 | 1088
  Other Histology | 2 | 3 | 5
Sites of Metastatic Disease [Number; unit: participants] — Participants may record multiple sites of metastatic disease.
  participants
    Bone | 120 | 131 | 251
    Brain | 28 | 30 | 58
    Liver | 109 | 117 | 226
    Lung | 453 | 453 | 906
    Lymph Nodes | 431 | 451 | 882
    Peritoneal | 20 | 17 | 37
    Pleural | 149 | 155 | 304
    Skin | 9 | 8 | 17
    Soft Tissue | 23 | 21 | 44
    Other | 156 | 146 | 302

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Time (OS)
Description: Overall survival is defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive. OS was estimated by the Kaplan-Meier method.
Time Frame: Randomization to Death from Any Cause (Up to 31 Months)
Population: All randomized participants. Censored participants: Necitumumab + Gemcitabine + Cisplatin = 127, Gemcitabine + Cisplatin = 106
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Necitumumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin
Number analyzed (Participants) | 545 | 548
Months | 11.5 [10.4 to 12.6] | 9.9 [8.9 to 11.1]
Statistical Analysis 1: Comparison: Necitumumab + Gemcitabine + Cisplatin vs Gemcitabine + Cisplatin; Test type: Superiority or Other; p = 0.0120, Log Rank; Hazard Ratio (HR) = 0.842, 95% CI 2-sided [0.736 to 0.962]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization until the first radiographic documentation of objective measured progressive disease as defined by RECIST (Version 1.0), or death from any cause. Progressive Disease (PD) was defined as having at least a 20% increase in the sum of the longest diameter of target lesions. Participants who die without a reported prior progression were considered to have progressed on the day of their death. Participants who did not progress or were lost to follow-up were censored at the day of their last radiographic tumor assessment. If no baseline or postbaseline radiologic assessment was available, the participants were censored at the date of randomization. If death or PD occurs after two or more consecutive missing radiographic visits, censoring occurred at the date of the last radiographic visit prior to the missed visits.
Time Frame: Randomization to Measured Progressive Disease or Death from Any Cause (Up to 31 Months)
Population: All randomized participants. Censored participants: Necitumumab + Gemcitabine + Cisplatin = 114, Gemcitabine + Cisplatin = 131
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Necitumumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin
Number analyzed (Participants) | 545 | 548
months | 5.7 [5.6 to 6.0] | 5.5 [4.8 to 5.6]
Statistical Analysis 1: Comparison: Necitumumab + Gemcitabine + Cisplatin vs Gemcitabine + Cisplatin; Test type: Superiority or Other; p = 0.0201, Log Rank; Hazard Ratio (HR) = 0.851, 95% CI 2-sided [0.743 to 0.975]

3. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR) (Objective Response Rate [ORR])
Description: ORR is confirmed best overall tumor response of CR or PR. According to RECIST v1.0, CR was defined as the disappearance of all target and non-target lesions. PR defined as a >=30% decrease in the sum of the longest diameters (LD) of the target lesions, taking as reference the baseline sum of the LD; Percentage of participants was calculated as: (total number of participants with CR or PR from start of the treatment until disease progression or recurrence)/total number of participants treated) * 100.
Time Frame: Baseline to Measured Progressive Disease (Up to 31 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Necitumumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin
Number analyzed (Participants) | 545 | 548
percentage of participants | 31.2 [27.4 to 35.2] | 28.8 [25.2 to 32.8]
Statistical Analysis 1: Comparison: Necitumumab + Gemcitabine + Cisplatin vs Gemcitabine + Cisplatin; Test type: Superiority or Other; p = 0.3997, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.86 to 1.45]

4. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF is defined as the time from the date of randomization until the date of the first radiographic documentation of PD, death from any cause, discontinuation of treatment for any reason, or initiation of new cancer therapy. Participants who withdrew from the study for reasons other than progression or death were censored at the date of study withdrawal. Participants who did not meet any of the criteria for treatment failure were censored at their date of last contact in the study.
Time Frame: Randomization to Measured Progressive Disease, Death From Any Cause, Discontinuation of Treatment or Initiation of New Anticancer Therapy (Up to 31 Months)
Population: All randomized participants. Censored participants: Necitumumab + Gemcitabine + Cisplatin = 16, Gemcitabine + Cisplatin =20
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Necitumumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin
Number analyzed (Participants) | 545 | 548
Months | 4.3 [4.2 to 4.8] | 3.6 [3.3 to 4.1]
Statistical Analysis 1: Comparison: Necitumumab + Gemcitabine + Cisplatin vs Gemcitabine + Cisplatin; Test type: Superiority or Other; p = 0.0061, Log Rank; Hazard Ratio (HR) = 0.844, 95% CI 2-sided [0.747 to 0.953]

5. Secondary Outcome: Mean Change From Baseline in Patient Reported Outcomes (PRO) Using the European Quality of Life-5 Dimension (EQ-5D)
Description: The EQ-5D is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a three level scale 1-3 (no problem, some problems, and major problems). These combinations of attributes were converted into a weighted health-state Index Score according to the United Kingdom (UK) population-based algorithm. The possible values for the Index Score ranged from -0.59 (severe problems in all 5 dimensions) to 1.0 (no problem in any dimension).
Time Frame: Baseline, Cycle 6 (Cycle = 3 Weeks)
Population: All randomized participants who had evaluable baseline and postbaseline EQ-5D data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Necitumumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin
Number analyzed (Participants) | 305 | 245
units on a scale | -0.0053 (0.23626) | -0.0083 (0.23866)

6. Secondary Outcome: Mean Change From Baseline in PRO Using the Outcomes Lung Cancer Symptom Scale (LCSS)
Description: The LCSS consisted of 9 items: 6 items focused on lung cancer symptoms [loss of appetite, fatigue, cough, dyspnea (shortness of breath), hemoptysis (blood in sputum), and pain] and 3 items were global items (symptom distress, interference with activity level, and global quality of life). Participant responses to each item were measured using visual analogue scales (VAS) with 100-mm lines. A higher score for any item represented a higher level of symptoms/problems. Scores for each of the reported categories ranged from 0 (for best outcome) to 100 (for worst outcome). The Average Symptom Burden Index (ASBI) was the mean of the 6 symptom items of the LCSS, and the Total LCSS was the mean of all 9 LCSS items. ASBI and Total LCSS were not computed for a participant if he/she had 1 or more missing values for the 6 and 9 items, respectively.
Time Frame: Baseline, Cycle 6 (Cycle = 3 Weeks)
Population: All randomized participants who had evaluable data for LCSS.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Necitumumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin
Number analyzed (Participants) | 545 | 548
millimeter (mm)
  Loss of Appetite (n=304, 242) | 1.8 (31.84) | 1.5 (29.30)
  Fatigue (n=302, 242) | 6.3 (29.15) | 3.5 (25.29)
  Cough (n=303, 243) | -7.8 (28.05) | -9.1 (25.74)
  Dyspnea (n=305, 244) | -2.8 (26.52) | -1.8 (25.27)
  Pain (n=302, 243) | -3.3 (17.98) | -2.2 (17.22)
  Overall Symptoms (n=303, 242) | -0.3 (26.19) | -0.6 (26.92)
  Interference (n=306,241) | 3.8 (29.74) | 2.2 (26.79)
  Quality of Life (n=305, 243) | -0.3 (27.35) | -1.6 (24.71)
  Average Symptom Burden Index (ASBI) (n=294, 234) | -1.9 (16.55) | -1.5 (16.52)
  LCSS Total Score (n=290, 228) | -0.8 (17.03) | -0.8 (16.17)

7. Secondary Outcome: Number of Participants With an Epidermal Growth Factor Hormone (EGFR) Protein Expression Measured by Immunohistochemistry (IHC)
Description: EGFR IHC Histoscore H-score = weighted sum of % 1+ cells, twice % 2+ cells, and three times % 3+ cells. IHC H-score criteria was used to assess participants with a low EGFR expression defined by a H-score cutoff value of <200 and participants with a high EGFR expression defined by a H-score of cutoff value of >=200.
Time Frame: 31 Months
Population: All randomized participants who received at least one dose of study drug and had evaluable data for EGFR IHC.
Measure: Number; unit: participants
Arm/Group | Necitumumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin
Number analyzed (Participants) | 486 | 496
participants
  0 | 24 | 23
  >0 | 462 | 473
  <200 | 295 | 313
  ≥200 | 191 | 183

8. Secondary Outcome: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Necitumumab
Time Frame: Day 1 of Cycle 2, 3, 4, 5 and 6 Prior to Necitumumab Drug Infusion, Up to 24 Months
Population: All randomized participants who received at least one dose of study drug and had evaluable data for PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (ug/mL)
Arm/Group | Necitumumab + Gemcitabine + Cisplatin
Number analyzed (Participants) | 545
micrograms/milliliter (ug/mL)
  Predose Cycle 2 Day 1 (n=419) | 52.4 (95.9)
  Predose Cycle3 Day 1 (n=386) | 76.6 (80.6)
  Predose Cycle 4 Day 1 (n=344) | 94.5 (92.2)
  Predose Cycle 5 Day 1 (n=297) | 101 (90)
  Predose Cycle 6 Day 1 (n=262) | 98.5 (80)

9. Secondary Outcome: Number of Participants With a Serum Anti-Necitumumab Antibody Assessment
Description: A participant was considered to have an anti-Necitumumab antibody response if anti-drug antibodies (ADA) were detected at any time point.
Time Frame: Baseline through 31 Months
Population: All randomized participants who received who received at least 1 dose of drug and had evaluable data for antibodies.
Measure: Number; unit: participants
Arm/Group | Necitumumab + Gemcitabine + Cisplatin
Number analyzed (Participants) | 528
participants
  Participants with at least 1 positive titer | 81
  Neutralizing antibody detected | 5

ADVERSE EVENTS:
Time Frame: Baseline Up To 156 Months
Description: All participants who received at least one dose of study drug. The adverse events were analyzed and reported according to the study treatments pre-specified in the statistical analysis plan.
Arm/Group | Necitumumab + Gemcitabine + Cisplatin | Gemcitabine + Cisplatin
All-Cause Mortality (participants affected / at risk) | 476/538 | 487/541
Serious Adverse Events (participants affected / at risk) | 262/538 | 208/541
Other Adverse Events (participants affected / at risk) | 518/538 | 512/541
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Necitumumab + Gemcitabine + Cisplatin (N=538) | Gemcitabine + Cisplatin (N=541)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 22 (22) | 17 (17)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (6) | 7 (7)
Leukopenia (Blood and lymphatic system disorders) | 6 (6) | 4 (4)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 20 (20) | 33 (33)
Pancytopenia (Blood and lymphatic system disorders) | 6 (6) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (17) | 20 (20)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 4 (4)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion malignant (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ototoxicity (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 5 (5)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 3 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 12 (12) | 2 (2)
Asthenia (General disorders) | 2 (2) | 3 (3)
Chills (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 8 (8) | 3 (3)
Fatigue (General disorders) | 3 (3) | 4 (4)
General physical health deterioration (General disorders) | 8 (8) | 7 (7)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 7 (7) | 4 (4)
Sudden death (General disorders) | 2 (2) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 6 (6) | 3 (3)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Dental gangrene (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Injection site abscess (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 4 (4)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 2 (2)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 13 (13) | 20 (20)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 2 (2) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 5 (5)
Septic shock (Infections and infestations) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection bacterial (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 12 (12) | 21 (21)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Underdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 6 (6) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Ecg signs of myocardial ischaemia (Investigations) | 0 (0) | 1 (1)
False positive investigation result (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 8 (8)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 6 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26 (26) | 23 (23)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 4 (4) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Radial nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 3 (3) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 4 (4) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 2 (2)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 5 (5)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 8 (8) | 6 (6)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 9 (9)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 9 (9)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Social stay hospitalisation (Social circumstances) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava occlusion (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Necitumumab + Gemcitabine + Cisplatin (N=538) | Gemcitabine + Cisplatin (N=541)
Anaemia (Blood and lymphatic system disorders) | 221 (221) | 246 (246)
Leukopenia (Blood and lymphatic system disorders) | 71 (71) | 85 (85)
Neutropenia (Blood and lymphatic system disorders) | 220 (220) | 229 (229)
Thrombocytopenia (Blood and lymphatic system disorders) | 103 (103) | 124 (124)
Abdominal pain upper (Gastrointestinal disorders) | 31 (31) | 29 (29)
Constipation (Gastrointestinal disorders) | 111 (111) | 101 (101)
Diarrhoea (Gastrointestinal disorders) | 84 (84) | 60 (60)
Dyspepsia (Gastrointestinal disorders) | 27 (27) | 22 (22)
Nausea (Gastrointestinal disorders) | 265 (265) | 284 (284)
Stomatitis (Gastrointestinal disorders) | 58 (58) | 32 (32)
Vomiting (Gastrointestinal disorders) | 153 (153) | 134 (134)
Asthenia (General disorders) | 125 (125) | 112 (112)
Fatigue (General disorders) | 117 (117) | 121 (121)
Oedema peripheral (General disorders) | 44 (44) | 42 (42)
Pyrexia (General disorders) | 70 (70) | 61 (61)
Paronychia (Infections and infestations) | 36 (36) | 1 (1)
Urinary tract infection (Infections and infestations) | 31 (31) | 13 (13)
Blood creatinine increased (Investigations) | 49 (49) | 41 (41)
Weight decreased (Investigations) | 73 (73) | 36 (36)
Decreased appetite (Metabolism and nutrition disorders) | 162 (162) | 153 (153)
Hyperglycaemia (Metabolism and nutrition disorders) | 28 (28) | 16 (16)
Hyperkalaemia (Metabolism and nutrition disorders) | 27 (27) | 19 (19)
Hypokalaemia (Metabolism and nutrition disorders) | 37 (37) | 27 (27)
Hypomagnesaemia (Metabolism and nutrition disorders) | 159 (159) | 82 (82)
Hyponatraemia (Metabolism and nutrition disorders) | 23 (23) | 29 (29)
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 (31) | 31 (31)
Back pain (Musculoskeletal and connective tissue disorders) | 38 (38) | 30 (30)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 (27) | 21 (21)
Dizziness (Nervous system disorders) | 55 (55) | 42 (42)
Headache (Nervous system disorders) | 57 (57) | 32 (32)
Insomnia (Psychiatric disorders) | 29 (29) | 30 (30)
Cough (Respiratory, thoracic and mediastinal disorders) | 93 (93) | 72 (72)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 93 (93) | 79 (79)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 40 (40) | 16 (16)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 49 (49) | 22 (22)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 29 (29) | 12 (12)
Acne (Skin and subcutaneous tissue disorders) | 47 (47) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 76 (76) | 70 (70)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 80 (80) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 35 (35) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 39 (39) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 252 (252) | 32 (32)
Skin fissures (Skin and subcutaneous tissue disorders) | 27 (27) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days